CLINICAL TRIAL: NCT02812784
Title: Can Nephrocheck™ Predict the Reversibility of Early, Acute Kidney Injury During Septic Shock?
Acronym: AKI-CHECK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2015_843_0022
Record Dates: First submitted 2016-06-20; First posted 2016-06-24 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Heading
Keywords: Nephrocheck™; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine blood

INTERVENTIONS:
Device: Nephrocheck TM

SUMMARY:
Patients with septic shock in the intensive care unit have an elevated risk of developing acute kidney injury (AKI).

DETAILED DESCRIPTION:
Patients with septic shock in the intensive care unit have an elevated risk of developing acute kidney injury (AKI). AKI is an independent factor for mortality. Interventions that limit the worsening of renal function might have an impact on the mortality rate in these patients. Given the absence of validated pharmacological treatments for limiting the progression of AKI or for accelerating recovery from AKI, early intervention and the restoration of the glomerular filtration rate (GFR) in this context of hemodynamic change during the initial phase of septic shock might improve the patients' prognosis. One major challenge is therefore how to determine whether or not the AKI is reversible. The best-studied biomarkers (NGAL and KIM 1) have little discriminant power in septic patients because of their poor specificity or unsuitable kinetics for very early diagnosis. The combination of urine assays for tissue inhibitor of metalloproteinase 2 (TIMP2) and insulin-like growth factor binding protein 7 (IGFBP7) has shown good diagnostic performance for the very early detection of the risk of developing AKI in the following 12 hrs. Urine levels of these two markers specifically reflect damage to kidney tubules. Moreover, the levels appear to be strongly correlated with the severity of tubule damage. Thus, one can reasonably hypothesize that measurement of these markers in the very early stages of septic shock might determine the presence and severity of kidney tubule damage. A threshold (yet to be defined) would help to differentiate between (i) transient, non-severe injury and (ii) injury that is already too severe to be reversible.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Septic shock (according to Bone's criteria) within 4 hours of introduction of catecholamines
* AKI, characterized by a KDIGO score ≥ 1
* Social security coverage

Exclusion Criteria:

* AKI requiring emergency RRT (in the critical care physician's opinion).
* Anuria
* Stage 4-5 chronic kidney failure with a GFR below 30 ml/min.
* Rapidly progressing renal disorders (glomerulonephritis, HUS, blockage, etc.)
* Obstructive AKI
* Probable glomerular damage (nephritic syndrome, nephrotic syndrome, chronic glomerulonephritis)
* Pregnancy or breastfeeding
* Legal guardianship or lack of social security coverage.
* Cardiocirculatory arrest
* Life expectancy <48 hours.
* Child C cirrhosis
* Prior occurrence of AKI during the current hospital stay
* Transplantation
* Subject participating in another study with an exclusion period ongoing at the time of the pre-inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Septic shock (according to Bone's criteria) within 4 hours of introduction of catecholamines
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2015-09-16 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
KDIGO classification | 72 hours
  predictive value of Nephrocheck™ with regard to the reversibility of AKI, defined as the recovery of normal renal function (KDIGO 0) in the 72 hours following inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Julien MAIZEL, MD, PhD, Principal Investigator — CHU Amiens
Locations (11):
- France (11):
  - CHU Amiens, Amiens
  - CH Avranches-Granville, Avranches
  - CH Cahors, Cahors
  - CH Dax, Dax
  - CH Marc Jacquet, Melun
  - CH de Mont-de-Marsan, Mont-de-Marsan
  - CHU Montpellier, Montpellier
  - CH Paris-Saint Joseph, Paris
  - CHU Poitiers, Poitiers
  - CHU Saint-Etienne, Saint-Etienne
  - CH Salon-de-provence, Salon-de-Provence

REFERENCES:
- [Derived] Titeca-Beauport D, Daubin D, Van Vong L, Belliard G, Bruel C, Alaya S, Chaoui K, Andrieu M, Rouquette-Vincenti I, Godde F, Pascal M, Diouf M, Vinsonneau C, Klouche K, Maizel J. Urine cell cycle arrest biomarkers distinguish poorly between transient and persistent AKI in early septic shock: a prospective, multicenter study. Crit Care. 2020 Jun 1;24(1):280. doi: 10.1186/s13054-020-02984-6. PMID 32487237